CLINICAL TRIAL: NCT06626256
Title: A Phase 1 Safety and Efficacy Study of STIL101 for Injection in Locally Advanced, Unresectable, or Metastatic Pancreatic Ductal Adenocarcinoma, Colorectal Cancer, Renal Cell Carcinoma, Cervical Cancer, and Melanoma
Brief Title: STIL101 for Injection for the Treatment of Locally Advanced, Metastatic or Unresectable Pancreatic Cancer, Colorectal Cancer, Renal Cell Cancer, Cervical Cancer and Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no resource
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24231; NCI-2024-08121 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24231 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Cervical Carcinoma; Locally Advanced Colorectal Carcinoma; Locally Advanced Malignant Solid Neoplasm; Locally Advanced Melanoma; Locally Advanced Pancreatic Ductal Adenocarcinoma; Locally Advanced Renal Cell Carcinoma; Metastatic Cervical Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Pancreatic Ductal Adenocarcinoma; Metastatic Renal Cell Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Cervical Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Unresectable Cervical Carcinoma; Unresectable Colorectal Carcinoma; Unresectable Malignant Solid Neoplasm; Unresectable Melanoma; Unresectable Pancreatic Ductal Adenocarcinoma; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis; Melanoma; Carcinoma, Renal Cell; Pancreatic Neoplasms | interventions — aldesleukin; Biopsy; Specimen Handling; Cyclophosphamide; fludarabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (STIL101 for injection) (Experimental): Patients undergo excisional biopsy and continue receiving standard of care therapy for 3-4 months prior to the start of study therapy. Patients with successful generation of STIL101 for injection receive cyclophosphamide IV over 2 hours on days -5 to -4, fludarabine IV over 30 minutes on days -5 to -1 and STIL101 for injection IV on day 0 in the absence of disease progression or unacceptable toxicity. Patients also receive aldesleukin SC QD on day 0 for up to 6-10 days. Additionally, patients undergo blood sample collection, biopsy, CT and optional MRI throughout the study.
  Interventions: Biological: Aldesleukin; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Excisional Biopsy; Drug: Fludarabine; Procedure: Magnetic Resonance Imaging; Procedure: Standard Treatment; Biological: Therapeutic Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Excisional Biopsy — Undergo excisional biopsy
  Other Names: Biopsy, Excisional; surgical biopsy
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Standard Treatment — Receive standard of care therapy
Biological: Therapeutic Tumor Infiltrating Lymphocytes — Given STIL101 for injection IV
  Other Names: Tumor Infiltrating Lymphocytes

SUMMARY:
This phase I trial tests the safety and side effects of STIL101 for injection and how well it works in treating patients with pancreatic cancer, colorectal cancer (CRC), renal cell cancer (RCC), cervical cancer (CC) and melanoma that has spread to nearby tissue or lymph nodes (locally advanced) or to other places in the body (metastatic) or that cannot be removed by surgery (unresectable). STIL101 for injection, an autologous (made from the patients own cells) cellular therapy, is made up of specialized white blood cells called lymphocytes or "T cells" collected from a piece of the patients tumor tissue. The T cells collected from the tumor are then grown in a laboratory to create STIL101 for injection. STIL101 for injection is then given to the patient where it may attack the tumor. Giving chemotherapy, such as cyclophosphamide and fludarabine, helps prepare the body to receive STIL101 for injection in a way that allows the T cells the best opportunity to attack the tumor. Aldesleukin is a form of interleukin-2, a cytokine made by leukocytes. Aldesleukin increases the activity and growth of white blood cells called T lymphocytes and B lymphocytes. Giving STIL101 for injection may be safe, tolerable and/or effective in treating patients with locally advanced, metastatic or unresectable pancreatic cancer, CRC, RCC, CC and melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the safety of administering STIL101 for injection in subjects with locally advanced, unresectable, or metastatic pancreatic ducal adenocarcinoma (PDAC), CRC, RCC CC or melanoma.

SECONDARY OBJECTIVES:

I. Summarize the efficacy observed due to STIL101 for injection in patients with locally advanced, unresectable or metastatic PDAC, CRC, RCC, CC or melanoma:

Ia. Overall response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and Immune-Modified (i)RECIST 1.0; Ib. Disease control rate (DCR) as measured from STIL101 infusion; Ic. Overall survival (OS) as measured from STIL101 infusion; Id. Progression-free survival (PFS) as measured from STIL101 infusion. II. Summarize pre-STIL101 for injection therapy and outcomes from first study-related procedure.

III. Evaluate the feasibility and timing of generating STIL101 for injection. IV. Describe STIL101 cell count in patients with respect to baseline characteristics, clinical outcome and adverse events.

EXPLORATORY OBJECTIVE:

I. Biological correlatives associated with STIL101 for injection creation and infusion.

OUTLINE:

Patients undergo excisional biopsy and continue receiving standard of care therapy for 3-4 months prior to the start of study therapy. Patients with successful generation of STIL101 for injection receive cyclophosphamide intravenously (IV) over 2 hours on days -5 to -4, fludarabine IV over 30 minutes on days -5 to -1 and STIL101 for injection IV on day 0 in the absence of disease progression or unacceptable toxicity. Patients also receive aldesleukin subcutaneously (SC) once daily (QD) on day 0 for up to 6-10 days. Additionally, patients undergo blood sample collection, biopsy, computed tomography (CT) and optional magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at days 42, 56, 70 and 84 then every 2-4 weeks up to week 96 or progression. Patients who discontinued treatment are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agree to research biopsies while on-study

  * Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening, while the request for a translated full consent is processed
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Anticipated life expectancy of > 6 months at the time of enrollment
* Participants with pancreatic ductal adenocarcinoma (PDAC), colorectal cancer (CC), renal cell carcinoma (RCC), cervical cancer (CC) and melanoma, meeting the following criteria will be eligible:

  * Cytologically or histologically confirmed locally advanced, unresectable, or metastatic PDAC, CRC, RCC, CC, melanoma
  * Patients must have received at least 1 line of standard therapy prior to receiving STIL101 for injection. Note: Patients may be enrolled prior to starting treatment to harvest tumor and blood samples for tumor infiltrating lymphocyte (TIL) generation
  * For pancreatic cancer patients:

    * Patients on first line treatment will need to receive at least 4 months of standard chemotherapy before receiving STIL101 for injection
    * In the second line setting, these patients may opt to receive STIL101 for injection at any time
  * For melanoma cancer patients: Patients need to have received prior PD1 therapy and BRAF inhibitor treatment in patients with a V600E mutation
  * For RCC, CRC, CC patients: Patients need to have failed at least 1 line of prior therapy
* Measurable disease by RECIST 1.1
* At least one lesion (or aggregate of lesions resected) that can be safety biopsied (excisional) and yield a volume (target of > 1cm^3) to generate STIL101 for injection (principal investigator [PI] discretion)
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3

  * NOTE: Growth factor is not permitted within 14 days of screening ANC assessment
* Platelets ≥ 100,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of screening platelet assessment
* Hemoglobin ≥ 8 g/dL

  * NOTE: Red blood cell transfusions are not permitted within 14 days of screening platelet assessment
* Total bilirubin ≤ 2 x upper limit of normal (ULN) (unless participant has Gilbert's disease which allows total bilirubin ≤ 3 x ULN)
* Aspartate aminotransferase (AST) ≤ 3 x ULN; ≤ 5.0 x ULN if hepatic metastases are present
* Alanine transaminase (ALT) ≤ 3 x ULN; ≤ 5.0 x ULN if hepatic metastases are present
* Creatinine clearance (CRCl) of ≥ 40 mL/min per 24-hour urine test or the Cockcroft-Gault formula
* Oxygen (O2) saturation > 92% on room air not requiring oxygen supplementation

  * Note: To be performed within 28 days prior to start of protocol therapy
* Left ventricular ejection fraction (LVEF) ≥ 50%

  * Note: To be performed within 8 weeks prior to start of protocol therapy
* If not receiving anticoagulants: International normalized ratio (INR) or prothrombin (PT) ≤ 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN. If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Seronegative for HIV antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), hepatitis B virus (HBV) (surface antigen negative), and syphilis (RPR)

  * If seropositive for HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetected
* QuantiFERON-TB Gold or equivalent

  * Results do not impact patient eligibility; however, the test must be initiated prior to enrollment
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior organ transplant
* Concomitant herbal medications with exception to cannabidiol (CBD), which is allowed
* Continuous systemic steroid therapy (i.e., > 10 mg/day of prednisone or other steroid equivalent dose) or other immunosuppressive therapies. Physical replacement doses (i.e., adrenocortical insufficiency), inhaled or topical steroids at ≤ 10 mg/day of prednisone or another steroid equivalent dose are permissible in the absence of active auto-immune disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents, including history of hypersensitivity to any drugs of the aminoglycoside group
* Prior or current known uveitis within 6 months of informed consent
* Active viral, bacterial, or fungal infection requiring treatment. Patients must be seronegative for the human immunodeficiency virus (HIV) and syphilis (RPR). Patients with hepatitis infections are allowed with undetected viral load
* Primary immunodeficiency (such as severe combined immunodeficiency [SCID] or acquired immunodeficiency syndrome [AIDS])
* End-stage renal disorder requiring hemodialysis
* Class III/IV cardiovascular disability according to the New York Heart Association (NYHA) Classification
* Known clinically significant pulmonary conditions within 6 months of informed consent
* Prior or concurrent malignancy. Prior malignancies with a low probability of recurrence requiring treatment such as the following are allowed: carcinoma in situ of the cervix, nonmelanoma skin cancer and low grade (Gleason score ≤ 6=Gleason group 1) localized prostate cancer. Prior malignancies not listed require PI approval
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Infusion limiting toxicities (ILTs) | From the start of STIL101 for injection up to 28 days
  Assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. ILTs will be summarized by severity, grade and attribution.
Treatment-related adverse events (AEs) | Up to 2 years
  Assessed by NCI CTCAE v 5.0. AEs will be summarized by severity, grade and attribution.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years
  The proportion of subjects with confirmed complete response (CR) / immune related (i)CR or partial response (PR) / iPR will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and Immune-Modified (i)RECIST 1.0.
Disease control rate | From start of STIL101 for injection infusion for at least one post-treatment scan up to 2 years
  The proportion of subjects who achieve CR/iCR, PR/iPR or maintain at least stable disease will be assessed using RECIST 1.1/iRECIST 1.0.
Overall survival | From the start of STIL101 for injection until death due to any cause up to 2 years
  Analysis will be descriptive.
Overall survival | From excisional biopsy until death due to any cause up to 2 years
  Analysis will be descriptive.
Progression-free survival | From start of STIL101 for injection infusion until documented progressive disease or death due to any cause up to 2 years
  Analysis will be descriptive.
Failure to receive STIL101 after excisional biopsy | Up to 2 years
  Analysis will be descriptive.
Time to lymphodepleting chemotherapy | From subject informed consent to start of lymphodepleting chemotherapy up to 2 years
  Analysis will be descriptive.
Excisional biopsy complication rate | Up to 2 years
  Analysis will be descriptive.
STIL101 for injection generation times | Up to 2 years
  Analysis will be descriptive.
Successful STIL101 for injection generation and administration | Up to 2 years
  Success rate for generation will be summarized and causes of failure will be documented. Those unable to receive STIL101 for injection will also be summarized.
STIL101 cell count | Up to 2 years
  STIL101 cell count in patients with respect to baseline characteristics, clinical outcome and AEs will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — City of Hope Medical Center